CLINICAL TRIAL: NCT04917224
Title: Phase II Study of LUNG Stereotactic Adaptive Ablative Radiotherapy for Central and Ultracentral Tumors
Brief Title: Study of LUNG Stereotactic Adaptive Ablative Radiotherapy
Acronym: LUNG STAAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ViewRay (funding agency) has filed under Chapter 11, U.S. Bankruptcy Code. ViewRay's clinical research support is paused and studies will not be paid directly by ViewRay. As such, the sponsor has closed the study without enrolling participants.
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KOT-005
Record Dates: First submitted 2021-05-11; First posted 2021-06-08 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer; Lung Tumor
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Central lung tumors (Experimental): Gross tumor volume (GTV) less than or equal to 1 cm from a lobar bronchus
  Interventions: Radiation: Stereotactic Adaptive Ablative Radiotherapy at 50 Gy (Gray)
- Cohort B: Ultra-central lung tumors (Experimental): Gross tumor volume (GTV) less than or equal to 1 cm from the mainstem bronchus, trachea, or esophagus
  Interventions: Radiation: Stereotactic Adaptive Ablative Radiotherapy at 60 Gy (Gray)

INTERVENTIONS:
Radiation: Stereotactic Adaptive Ablative Radiotherapy at 50 Gy (Gray) — Cohort A will include 30 patients with central tumors; the dose regimen prescribed is 50 Gy (Gray) in 5 fractions with a 40 hour inter-fraction interval.
  Arms: Cohort A: Central lung tumors
Radiation: Stereotactic Adaptive Ablative Radiotherapy at 60 Gy (Gray) — Cohort B will include 30 patients with ultra-central tumors; the dose regimen prescribed is 60 Gy (Gray) in 8 fractions on consecutive days.
  Arms: Cohort B: Ultra-central lung tumors

SUMMARY:
The proposed study expands on the principles of SBRT (Stereotactic Body Radiation Therapy) and SABR (Stereotactic Ablative Radiotherapy) for centrally located NSCLC (Non-Small Cell Lung Cancer) to further optimize outcomes in this patient population with utilization of the adaptive workflow to maintain tumor control rates but decrease the incidence and grade of treatment-related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Clinical diagnosis of NSCLC
* Stage T1-2b (≤ 5 cm)

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year (i.e., carcinomas in situ of the breast, oral cavity, or cervix are permissible); previous lung cancer, if the patient is disease-free for a minimum of 1 year is permitted;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Prior chemotherapy for the study cancer
* Plans for the patient to receive other local therapy (including standard fractionated radiotherapy and/or surgery) while on this study, except at disease progression
* Plans for the patient to receive systemic therapy (including standard chemotherapy or biologic targeted agents), while on this study, except at disease progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2031-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Treatment completion | Plus or minus 5 days of treatment
  Number of patients who completed treatment within +/- 5 days of intended treatment.
Number of patients experiencing adverse events | 12-month of treatment
  No greater than 15 percent of patients experience a 12-month ≥ grade 3 toxicity and ≤1 grade 5 toxicity possibly, probably, or definitely related to treatment.

SECONDARY OUTCOMES:
Primary Tumor Control Rate | 1 year of treatment
  Primary tumor control rate at the maximum tolerated dose (MTD) based on each treatment cohort.
Progression-free survival (PFS) | 1 year of treatment
  Progression-free survival (PFS) is defined as the first occurrence of local and/or regional disease progression, distant metastases, second primary tumor, or death due to any cause. PFS time is measured from the date of start of SBRT to the date of the failure event for PFS.
Overall survival (OS) | 1 year of treatment
  Overall survival (OS) time is measured from the date of start of SBRT to the date of death due to any cause.
Functional Assessment of Cancer Therapy - Lung (FACT-L) | Baseline
  The Functional Assessment of Cancer Therapy - Lung (FACT-L) quality of life instrument has been extensively used for measuring quality of life in patients with lung cancer. There are 5 sections dealing with physical, family, emotional, functional well-being, and additional concerns. There are nine questions that are specific to lung cancer (LSC), including shortness of breath, cough, etc. The TOI (Trial Outcome Index) is the sum of the scores on the LCS and the physical well-being and functional well-being subscales of the FACT-L scale.
EQ-5D-5L | 3 and 12-month follow-up
  The five-item index score from EQ-5D-5L will be used to generate utility scores that will lie between 0 (Worst health state) and 1 (Best health state).
Late-Toxicity | 1 year of treatment
  Rate of late (>1 year) ≥ grade 3 adverse events related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh Kotecha, MD, Principal Investigator — Miami Cancer Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenberg SA, Mak R, Kotecha R, Loo BW Jr, Senan S. The Nordic-HILUS Trial: Ultracentral Lung Stereotactic Ablative Radiotherapy and a Narrow Therapeutic Window. J Thorac Oncol. 2021 Oct;16(10):e79-e80. doi: 10.1016/j.jtho.2021.06.030. No abstract available. PMID 34561039
- See also: Related Info — https://baptisthealth.net/en